CLINICAL TRIAL: NCT06849882
Title: Dubousset Functional Test: an Investigation of Its Validity and Reliability in Individuals with Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: Inonu University (Other)
Collaborators: Kayseri Erciyes University Faculty of Medicine (Unknown)
Responsible Party: Principal Investigator, Betul Ergun, RESEARCH ASSISTANT, TC Erciyes University
Other Study IDs: Dubousset -MS
Record Dates: First submitted 2025-02-17; First posted 2025-02-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: MS (Multiple Sclerosis)
Keywords: Multiple Sclerosis; Dubousset Functional Test; Validity; Reliability
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — samples will not be stored and DNA will not be used within the scope of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dubousset Functional Test: Individuals with Multiple Sclerosis

SUMMARY:
Multiple sclerosis (MS) is an autoimmune disease characterized by neuroinflammation and neurodegeneration in the central nervous system. The disease affects the white matter, cortex and deep gray matter of the central nervous system and is characterized by inflammatory-demyelinating lesions and neuronal/axonal degeneration. Demyelination associated with these lesions and the accompanying axonal degeneration are responsible for neurological disability in MS. There are many scales and mobility and functional performance tests in the literature to assess balance, such as the Sit Reach Test, Timed Up and Go (TUG) test, Tinetti Performance Oriented Mobility Assessment (POMA), Berg Balance Scale (BBS) (5) and Balance Evaluation System Test (BESTest). The most appropriate balance assessment scales for individuals with MS are those that assess static and dynamic sitting balance while standing and dynamic balance only. Since balance in individuals with MS is a dynamic process that changes gradually, new measurement methods that can record these changes and determine the appropriate treatment for these variables are needed.

The Dubousset Functional Test (DFT) was developed by Dr. Jean Dubousset as a four-component practical assessment to evaluate the physical function and balance capacity of individuals with spinal deformity. The DFT consists of four components: getting up from an armless chair and walking 5 meters forward and backward, ascending and descending steps, transition from standing to sitting position, and gait assessment with a dual task test (counting backwards from 50). The difference of this test from the others is that it evaluates the spinopelvic muscle groups that are directly related to functionality, maintains the global trunk alignment of the individual and provides objective results about functional performance and balance. In addition, unlike other functional performance tests, the DFT assesses the neurophysiological effects of the process that requires individuals to perform two tasks at the same time by measuring their coordination, balance, attention and thinking skills during functioning through a dual task component. The validity and reliability of this test has been previously investigated in low back pain, stroke, parkinson's disease, elderly individuals and hemiplegia. In this study, it was aimed to examine the validity and reliability of the Dubousset functional test in individuals with multiple sclerosis.

DETAILED DESCRIPTION:
Socio-demographic characteristics, physical characteristics (age, body weight, height), educational status, occupation, duration of MS, age at onset of MS, clinical type of MS, number and site of attacks, presence of optic neuritis, EDSS score, medications, chronic diseases, and smoking will be recorded.

Expanded Disability Status Scale (EDSS): All volunteers participating in the study will undergo a neurologic examination and the disability rate will be evaluated using the EDSS for each individual with MS. The EDSS is scored between 0 and 10, with higher scores indicating more disability. A score of zero indicates completely normal functioning, while a score of 10 indicates death due to MS. Individuals with a score of 3.5 and below will be included in the study.

Test Procedures Demographic data will be recorded at the baseline assessment. Our study will be conducted in a "test-retest" design and the psychometric properties of the Dubousset Function Test (DFT) will be examined in individuals with MS. The DFT, TUG, dual-task TUG, Tinetti Performance Oriented Mobility Assessment (POMA), Berg Balance Scale (BBS), Functional Reach Test and 3-meter backward walking test (3MBWT) will be administered to individuals. The completion times of the DFT will be performed by the same physiotherapist. The second assessment (retest) will be performed 7 days after the first assessment (test) by the same physiotherapist to determine the reliability of the DFT. Rest periods of 2 minutes will be given between assessments to minimize the effects of fatigue. Participants will not receive any treatment for 7 days and the test-retest will be performed at the same time.

Dubousset Functional Test (DFT):

A conceptual four-component global functional assessment test - Dubousset Functional Test (DFT) will be applied to objectively measure the functional capacity of individuals (11). These four components are as follows;

1. Get Up and Walk Test: Individuals with MS will stand up unassisted from a seated position in a chair without arms, walk 5 meters (500 cm), turn around, walk back 5 meters and sit down again unassisted.
2. Step Test: individuals with MS will climb three steps of stairs from a starting position 50 cm away, turn around on the third step and walk back down.
3. Sit and stand test: Individuals with MS will sit on the floor from a standing position with assistance if necessary and stand up again with assistance if necessary.
4. Dual Task Test: Individuals with MS will walk 5 meters forward, turn around and walk 5 meters backward while performing a memory exercise (counting down from 50 in 2 intervals).

TUG (Timed Up and Go) Test: The TUG test is a tool designed to assess dynamic balance, walking speed and mobility. To complete the test, participants are required to get up from a chair with armrests, walk 3 m, turn, walk back and sit on the chair. The completion time of the test is recorded with a stopwatch (3).

Dual Task TUG (Additional Cognitive Task): During the TUG test, counting backwards by twos from 50 will be used as an additional cognitive task. When the test had to be repeated, individuals continued counting from the number they had left off. Counting errors will be ignored (12).

Tinetti POMA: It is also called the Tinetti Mobility Test and is a reliable and valid clinical test used to measure balance and walking abilities. It consists of a total POMA scale (POMA-T), a balance subscale (POMA-B) and a gait subscale (POMA-G). Each step is scored between 0 (maximum inability) and 2 (complete independence) (13).

Berg Balance Scale (BBS): It is a widely used measurement tool to assess functional balance. The BBS consists of 14 items and each item is scored between 0 and 4 according to the level of balance impairment. Higher scores on the BDI indicate better balance performance (14).

3 Meter Backward Walking Test (3MBWT): A distance of 3 meters (m) is measured and marked with black tape. Patients are asked to follow the black tape with their heels. When the "Start" command is given, they are asked to walk backwards quickly. When a distance of 3 meters is completed, they are told to stop (15).

Functional Reach Test (FRT) : It is a test that evaluates dynamic bilateral postural balance. At the beginning of the test, the dominant arm is placed in a 90° flexion position and the distance between the feet is set to 10 cm. The maximum distance a person can extend their arm horizontally forward without moving their feet is measured in centimeters. The maximum distance he/she can reach and return to the starting position without losing balance is recorded. The test will be repeated three times and the average of these three values will be taken (16).

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MS,
* Over 18 years of age and under 65 years of age,
* To be able to balance independently in standing position.
* EDSS score of 3.5 and below
* At the appropriate cognitive level to adapt to the tests to be performed in the study,
* Completed primary school level,

Exclusion Criteria:

* Relapse within the last 30 days,
* Loss of balance or gait disturbance affected by a condition other than MS,
* Being pregnant for female individuals,
* An attack of optic neuritis in the last month
* Individuals who are unable to perform the task due to sensory, cognitive or other problems will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty-three individuals with MS who met the inclusion criteria will be included in the study. G-Power 3.1.9.2 program was used to estimate the required sample size and it was observed that the effect obtained in the reference study was strong (d = 0.731) (17). As a result of the power analysis performed with the assumption that this effect size could be obtained again, it was calculated that 95% statistical power would be obtained at 95% confidence level if at least 33 people were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Dubousset Functional Testing in Individuals with MS | Day 1
  The aim of this study is to investigate the validity and reliability of the Dubousset functional test in individuals with multiple sclerosis.The Dubousset Functional Test consists of four components;
  1. Get Up and Walk Test: Individuals with MS will stand up unassisted from a seated position in a chair without arms, walk 5 meters (500 cm), turn around, walk back 5 meters and sit down again unassisted.
  2. Step Test: individuals with MS will climb three steps of stairs from a starting position 50 cm away, turn around on the third step and walk back down.
  3. Sit and stand test: Individuals with MS will sit on the floor from a standing position with assistance if necessary and stand up again with assistance if necessary.
  4. Dual Task Test: Individuals with MS will walk 5 meters forward, turn around and walk 5 meters backward while performing a memory exercise (counting down from 50 in 2 intervals).

SECONDARY OUTCOMES:
TUG (Timed Up and Go) Test | Day 1
  The TUG test is a tool designed to assess dynamic balance, walking speed and mobility. To complete the test, participants are required to get up from a chair with armrests, walk 3 m, turn, walk back and sit on the chair. The completion time of the test is recorded with a stopwatch (3).
Dual Task TUG (Additional Cognitive Task) | Day 1
  During the TUG test, counting backwards by twos from 50 will be used as an additional cognitive task. When the test had to be repeated, individuals continued counting from the number they had left off. Counting errors will be ignored.
Tinetti POMA | Day 1
  It is also called the Tinetti Mobility Test and is a reliable and valid clinical test used to measure balance and walking abilities. It consists of a total POMA scale (POMA-T), a balance subscale (POMA-B) and a gait subscale (POMA-G). Each step is scored between 0 (maximum inability) and 2 (complete independence).
Berg Balance Scale (BBS) | Day 1
  It is a widely used measurement tool to assess functional balance. The BBS consists of 14 items and each item is scored between 0 and 4 according to the level of balance impairment. Higher scores on the BDI indicate better balance performance.
3 Meter Backward Walking Test (3MBWT) | Day 1
  A distance of 3 meters (m) is measured and marked with black tape. Patients are asked to follow the black tape with their heels. When the "Start" command is given, they are asked to walk backwards quickly. When the 3-meter distance is completed, they are told to stop.
Functional Reach Test (FRT) | Day 1
  : It is a test that evaluates dynamic bilateral postural balance. At the beginning of the test, the dominant arm is placed in a 90° flexion position and the distance between the feet is set to 10 cm. The maximum distance a person can extend their arm horizontally forward without moving their feet is measured in centimeters. The maximum distance he/she can reach and return to the starting position without losing balance is recorded. The test will be repeated three times and the average of these three values will be taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided